CLINICAL TRIAL: NCT03846154
Title: Reintegrating Children Living at Landfills in Burundi Into Society by Means of a Comprehensive Family Program Addressing Maltreatment and Trauma-related Mental Health Symptoms
Brief Title: Reintegrating Children Living at Landfills in Burundi Into Society by Means of a Comprehensive Family Program Addressing Maltreatment and Mental Health Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Vivo international e.V. (Industry); Psychologues sans Frontières Burundi (Other); Université Lumière de Bujumbura (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Principal investigator, University of Konstanz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCR18
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Posttraumatic Stress Disorder; Aggressive Behaviour; Parental Maltreatment; Days Spent at the Landfill
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Children and adolescents in the intervention group received:
  1. A group intervention once a week for about 20 weeks, including psychoeducation on mental health and drug abuse, anger management, roles within families, developing plans for the future, communication skills, sex education.
  2. Access to schools and school material
  3. Family visits
  4. Their parents received training regarding agriculture and microcredit projects, and financial assistance
  5. FORNET if affected by trauma-related symptoms, and/or acting aggressive
  6. If needed medical assistance is provided
  7. If needed legal assistance is provided
  Interventions: Behavioral: Comprehensive family intervention including individual sessions of FORNET
- Control group (No Intervention): The control group was invited to participate in three interviews getting small amounts of money (~2,5 €) as decompensation of their time.

INTERVENTIONS:
Behavioral: Comprehensive family intervention including individual sessions of FORNET — 1. A group intervention once a week for about 20 weeks, including psychoeducation on mental health and drug abuse, anger management, roles within families, developing plans for the future, communication skills, sex education.
  2. Access to schools and school material
  3. Family visits
  4. Their parents received training regarding agriculture and microcredit projects, and financial assistance
  5. FORNET if affected by trauma-related symptoms, and/or acting aggressive
  6. If needed medical assistance /.) If needed, legal assistance
  Arms: Intervention group

SUMMARY:
Children living at the landfills of Bujumbura are often exposed to maltreatment, including emotional neglect and physical abuse, and traumatic experiences. Furthermore, they grow up in severe poverty. Addressing trauma-related mental health issues and aggressive behaviour by Narrative Exposure Therapy (FORNET), familial communication by family visits, interaction difficulties of children by a group intervention, poverty by financial support and economic training for mothers, medical problems by medical assistance, legal conflicts by legal advice, and providing access to school, we aimed at reintegrating those children within the Burundian school system and improving familial relationships.

The investigators want to provide evidence, that mental health interventions are an integral part of assisting children and families affected by poverty and violence.

ELIGIBILITY:
Inclusion Criteria:

* Spending days at the landfills of Bujumbura

Exclusion Criteria:

* Psychotic symptoms

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change of load of traumatic symptoms measured via the University of California at Los Angeles Posttraumatic Stress Disorder Reaction Index (scale administered by Clinicians) | baseline; 5 months follow-up; 9 months follow-up
  27 items assessing PTSD, 4 additional items assessing dissociation on a scale from 0 - 4. Due to scoring rules, total sum score ranges from 0 to 80; sub scale intrusion: 0 - 20; sub scale avoidance: 0 - 8; sub scale negative cognitions: 0 - 28; sub scale hyperarousal: 0 - 24; higher values indicate more severe PTSD symptoms; all items are summed up for the total score
Change of number of aggressive acts measured via an adaption of the Domestic and Community Violence Checklist | baseline; 5 months follow-up; 9 months follow-up
  32 items; answer categories: yes or no; sum score ranges from 0 - 32
Change of experienced parental maltreatment measured via a shortened version of the Maltreatment and Abuse Chronology of Exposure (MACE) | baseline; 5 months follow-up; 9 months follow-up
  total sum score ranges from 0 - 100; sum score of each sub scale ranges from 0 - 10
Change of number of days spent at the landfill | baseline; 5 months follow-up; 9 months follow-up
  during the last 14 days; sum ranges from 0 - 14

CONTACTS AND LOCATIONS:
Locations (1):
- vivo international & Psychologues sans Frontières mental health center, Bujumbura, Bujumbura Mairie Province, Burundi

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share IPD with other researchers not related to the institutions conducting the study. If data is shared, the PI will supervise those analysing the date, e.g., students writing their theses